CLINICAL TRIAL: NCT02829112
Title: Shulman Fasciitis Prevalence Study in Alsace
Acronym: SHULMAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6177
Record Dates: First submitted 2016-06-16; First posted 2016-07-12 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Shulman Fasciitis
Keywords: Shulman; fasciitis; Shulman fasciitis; eosinophilic fasciitis; inflammatory disease; prevalence
MeSH Terms: conditions — Fasciitis; Eosinophilic Fasciitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Shulman fasciitis or eosinophilic fasciitis (EF) is a rare inflammatory disease, usually benign but disabling, described by Shulman in 1974. The diagnosis is suggested by the clinic, confirmed by MRI and confirmed by histology, there really no published diagnostic criteria validated for this rare disease. The low number of cases reported in the literature reflects the difficulty of studying the epidemiology of this disease, to establish and evaluate therapeutic strategies and to assess prognosis. Work on this subject are few. To our knowledge, no study has previously used to estimate the incidence and prevalence of this disease. Therefore, the investigators want to determine the prevalence of FEs in Alsace in 2016 by a study "capture-recapture" using several independent sources of identification of cases in order to have recent epidemiological data and learn more about this disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Patients suffering from fasciitis Shulmande and living in Alsace at 1 January 2016

Exclusion Criteria:

* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients suffering from fasciitis Shulmande and living in Alsace at 1 January 2016
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Estimation of the prevalence of Shulman fasciitis in Alsace, the calculation will be carried out using the numerator of all the cases identified and in the denominator the general population (Alsatian population of both sexes) | all living patients in Alsace from 1 January 2016 to december 2016

CONTACTS AND LOCATIONS:
Locations (1):
- Service de rhumatologie, Les Hôpitaux Universitaires de Strasbourg, Centre national de référence " des maladies auto-immunes rares ", Strasbourg, France

IPD SHARING:
Plan to Share IPD: No